CLINICAL TRIAL: NCT05112328
Title: The Effects of Pancreatic Enzyme Supplementation in Critically Ill Patients on Enteral Feeding: Prospective Randomized Controlled Trial
Brief Title: The Effects of Pancreatic Enzyme Supplementation in Critically Ill Patients on Enteral Feeding
Acronym: PREZENT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Seung-Young Oh, Clinical Assistant Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2008-185-1153
Record Dates: First submitted 2021-10-07; First posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Critically Ill; Enteral Feeding; Exocrine Pancreatic Insufficiency
MeSH Terms: conditions — Critical Illness; Exocrine Pancreatic Insufficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Exocrine Pacancreatic enzyme(Norzyme Capsule 40000 capsules) after meals 3 times a day
  Interventions: Drug: Exocrine Pancreatic Enzyme
- Control (Placebo Comparator): Placebo after meals 3 times a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Exocrine Pancreatic Enzyme — Pancreatic enzyme supplementation for critically ill patients on enteral nutrition
  Other Names: Norzyme
  Arms: Intervention
Drug: Placebo — Placebo of Pancreatic enzyme for critically ill patients on enteral nutrition
  Arms: Control

SUMMARY:
Determine the effect of high-dose pancreatic enzyme supplementation on nutritional indicators and clinical course in critically ill patients undergoing enteral nutrition.

ELIGIBILITY:
Inclusion Criteria:

* Adults 19 years and older
* Hospitalized in the surgical/medical intensive care unit of the Seoul National University Hospital
* Enteral nutrition
* Patients who consented to this study
* Patients with risk factors for pancreatic exocrine dysfunction

  * Shock (Norepinephrine)
  * Sepsis (3 rd definition of sepsis)
  * Diabetes
  * Cardiac arrest
  * hyperlactatemia serum lactate > 2 mmol/L)
  * Mechanical ventilation
  * Continuous renal replacement therapy

Exclusion Criteria:

* chronic pancreatitis
* unresectable pancreatic cancer
* History of pancreatectomy
* Underlying diseases in which the effect of Exocrine pancreatic enzyme administration is difficult to show

  * Inflammatory bowel disease
  * Short bowel syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2021-07-07 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change of Phase angle (°) | Baseline, 7 days after starting enteral nutrition, 14 days after starting enteral nutrition
  Change from Baseline Phase angle (°) at 2 weeks or discharge

SECONDARY OUTCOMES:
Skeletal Muscle Mass (SMM) (kg) | Baseline, 7 days after starting enteral nutrition, 14 days after starting enteral nutrition
  Skeletal Muscle Mass (SMM) (kg)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Jongno-gu, South Korea